CLINICAL TRIAL: NCT06370442
Title: Intranasal Dexmedetomidine vs. Standard of Care for Emergency Department (ED) Procedural Sedation in the Older Adult
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Jay Brenner, Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2137695
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Altered Mental Status
Keywords: Sedation
MeSH Terms: interventions — Dexmedetomidine; Lorazepam; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lorazepam (Active Comparator)
  Interventions: Drug: Lorazepam
- Haloperidol (Active Comparator)
  Interventions: Drug: Haloperidol
- IN Dex (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine, 100mcg
  Other Names: Precedex
  Arms: IN Dex
Drug: Lorazepam — 0.5mg IV
  Other Names: Ativan
  Arms: Lorazepam
Drug: Haloperidol — 0.5mg IV
  Other Names: Haldol
  Arms: Haloperidol

SUMMARY:
The purpose of the study is to determine if intranasal dexmedetomidine could be an alternative to the current standard of care (injectable benzodiazepines or antipsychotics) for sedation prior to computerized tomography (CT) or magnetic resonance imaging (MRI) in those greater than or equal to 65 years of age (older adults) that are seen in the Emergency Department (ED).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Patients in need of sedation prior to either a computerized tomography (CT) or magnetic resonance imaging (MRI)

Exclusion Criteria:

* Patients who weigh < 50 kg
* Cardiac arrhythmias or QTc >450
* Intravenous access not standard of care or unable to obtain
* Patients with any allergies or contraindications to dexmedetomidine, haloperidol (i.e. patients diagnosed with Parkinson's) or lorazepam
* Patients with low blood pressure, defined as a less than 100/60 mmHg
* Patients with bradycardia (Heart rate < 60 bpm)
* Patients presenting with chief complaint of respiratory distress/failure
* Intranasal administration contradictions: nasal septal abnormalities, nasal trauma, epistaxis, excessive nasal mucus or blood, and intranasal damage, recent use of nasally administered vasoconstrictors such as cocaine, oxymetazoline, and phenylephrine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Sedation | Within one hour of administration
  The primary outcome is to determine if intranasal dexmedetomidine is as effective in producing moderate sedation on the Modified Observer's Assessment of Alertness/Sedation Scale (MOAAS) as standard of care intravenous medications in older adults. The minimum value on the Modified Observer's Assessment of Alertness/Sedation Scale is 0 and the maximum value is 5. Lower scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: William Paolo, MD, Study Chair — State University of New York - Upstate Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennedy M, Koehl J, Gao J, Ciampa KA, Hayes BD, Camargo CA Jr. Use of antipsychotic and sedative medications in older patients in the emergency department. J Am Geriatr Soc. 2022 Mar;70(3):731-742. doi: 10.1111/jgs.17590. Epub 2021 Nov 25. PMID 34820831
- [Result] Tobias JD, Leder M. Procedural sedation: A review of sedative agents, monitoring, and management of complications. Saudi J Anaesth. 2011 Oct;5(4):395-410. doi: 10.4103/1658-354X.87270. PMID 22144928
- [Result] Kienitz R, Kay L, Beuchat I, Gelhard S, von Brauchitsch S, Mann C, Lucaciu A, Schafer JH, Siebenbrodt K, Zollner JP, Schubert-Bast S, Rosenow F, Strzelczyk A, Willems LM. Benzodiazepines in the Management of Seizures and Status Epilepticus: A Review of Routes of Delivery, Pharmacokinetics, Efficacy, and Tolerability. CNS Drugs. 2022 Sep;36(9):951-975. doi: 10.1007/s40263-022-00940-2. Epub 2022 Aug 16. PMID 35971024
- [Result] Amore M, D'Andrea M, Fagiolini A. Treatment of Agitation With Lorazepam in Clinical Practice: A Systematic Review. Front Psychiatry. 2021 Feb 22;12:628965. doi: 10.3389/fpsyt.2021.628965. eCollection 2021. PMID 33692709
- [Result] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Result] Baumgartner K, Groff V, Yaeger LH, Fuller BM. The use of dexmedetomidine in the emergency department: A systematic review. Acad Emerg Med. 2023 Mar;30(3):196-208. doi: 10.1111/acem.14636. Epub 2022 Dec 19. PMID 36448276
- [Result] Barends CRM, Driesens MK, Struys MMRF, Visser A, Absalom AR. Intranasal dexmedetomidine in elderly subjects with or without beta blockade: a randomised double-blind single-ascending-dose cohort study. Br J Anaesth. 2020 Apr;124(4):411-419. doi: 10.1016/j.bja.2019.12.025. Epub 2020 Feb 3. PMID 32029262
- [Result] Pastis NJ, Hill NT, Yarmus LB, Schippers F, Imre M, Sohngen W, Randall O, Callahan SP, Silvestri GA. Correlation of Vital Signs and Depth of Sedation by Modified Observer's Assessment of Alertness and Sedation (MOAA/S) Scale in Bronchoscopy. J Bronchology Interv Pulmonol. 2022 Jan 1;29(1):54-61. doi: 10.1097/LBR.0000000000000784. PMID 34238838
- [Result] Uusalo P, Seppanen SM, Jarvisalo MJ. Feasibility of Intranasal Dexmedetomidine in Treatment of Postoperative Restlessness, Agitation, and Pain in Geriatric Orthopedic Patients. Drugs Aging. 2021 May;38(5):441-450. doi: 10.1007/s40266-021-00846-6. Epub 2021 Mar 16. PMID 33728561
- [Result] Gupta A, Dalvi NP, Tendolkar BA. Comparison between intranasal dexmedetomidine and intranasal midazolam as premedication for brain magnetic resonance imaging in pediatric patients: A prospective randomized double blind trial. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):236-240. doi: 10.4103/joacp.JOACP_204_16. PMID 28781452
- [Result] Sinnott J, Holthaus CV, Ablordeppey E, Wessman BT, Roberts BW, Fuller BM. The Use of Dexmedetomidine in the Emergency Department: A Cohort Study. West J Emerg Med. 2021 Aug 22;22(5):1202-1209. doi: 10.5811/westjem.2021.4.50917. PMID 34546899